CLINICAL TRIAL: NCT05417880
Title: Vitamin D, K2 Plus Empagliflozin Combination in Type Two Diabetes Mellitus
Acronym: VETA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Scotmann Pharmaceuticals (Industry)
Collaborators: University of Health Sciences Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VETAtrial
Record Dates: First submitted 2022-06-07; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Empagliflozin; Vitamin D3; Vitamin K2
MeSH Terms: conditions — Diabetes Mellitus | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Prospective Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Control group) (Active Comparator): Continue with current oral anti-hyperglycemic regime
  Interventions: Drug: Oral Hypoglycemic Agents,Oral
- Group 2 (Voreta group) (Active Comparator): Empagliflozin 10 mg OD
  Interventions: Drug: Voreta
- Group 3 ( Voreta + SunnyD PRO group ) (Experimental): Empagliflozin 10 mg OD + Vitamin D3 (2000 IU) + Vitamin K2 (100 mcg)
  Interventions: Drug: Voreta plus SunnyD PRO

INTERVENTIONS:
Drug: Oral Hypoglycemic Agents,Oral — Control group with routine current oral hypoglycemic agents for 3-6 months
  Other Names: Control group
  Arms: Group 1 (Control group)
Drug: Voreta — Empagliflozin 10 mg oral tablets Once Daily for 3-6 months
  Other Names: Voreta group
  Arms: Group 2 (Voreta group)
Drug: Voreta plus SunnyD PRO — Empagliflozin 10 mg oral tablets + Vitamin D3 ( 2000 IU ) + Vitamin K2 ( 100 mcg) Once Daily for 3-6 months
  Other Names: Voreta and SunnyD PRO group
  Arms: Group 3 ( Voreta + SunnyD PRO group )

SUMMARY:
The main purpose of the VETA trial is to verify the potential beneficial effects of the combination of micronutrients namely Vitamin D3 and K2 in combination with oral antihyperglycemic Empagliflozin in Diabetes Mellitus

DETAILED DESCRIPTION:
Empagliflozin:

Generally, Sodium-glucose co-transporter-2 inhibitors (SGLT2i), have important benefits for older people, such as a low risk of hypoglycemia, reduction of cardiovascular and renal risk, and an insulin-independent mechanism, allowing its use in disease of any duration. Advantages include lack of hypoglycemia as a side effect, and mild reduction in blood pressure and body weight.

The SGLT2i class is well-tolerated, though some caution is also suggested, including adjustment of concomitant therapies, such as insulin and antihypertensives, especially loop diuretics.

The 2022 latest guidelines by the American Diabetes Association recommend that if insulin is used in adults with type 2 diabetes, it is recommended that, for better efficacy and durability of treatment effect, combination therapy be employed using a glucagonlike peptide 1 receptor agonist and consideration may be given to combined therapy employing a sodium-glucose cotransporter 2 inhibitor and a glucagon-like peptide 1 receptor agonist, both with demonstrated cardiovascular benefit, "for additive reduction in the risk of adverse cardiovascular and kidney events" in patients "with type 2 diabetes and established atherosclerotic cardiovascular disease or multiple risk factors for atherosclerotic cardiovascular disease". Moreover, among patients with type 2 diabetes who have established atherosclerotic cardiovascular disease (ASCVD), sodiumglucose cotransporter-2 (SGLT2) inhibitors or glucacon-like peptide 1 (GLP-1) receptor agonists with proven cardiovascular benefit are recommended as part of glycemic management. The same guidelines recommend that among patients with ASCVD in whom heart failure coexists or is of special concern, SGLT2 inhibitors are recommended and patients who are unable to maintain glycemic targets on basal insulin in combination with oral medications can have treatment intensified with GLP-1 receptor agonists, SGLT2 inhibitors, or prandial insulin.

Conclusively, it is recommended that a sodium-glucose cotransporter-2 (SGLT2) inhibitor or glucagonlike peptide-1 receptor agonist (GLP-1 RA) with demonstrated cardiovascular disease benefit be administered to patients with type 2 diabetes who have established atherosclerotic cardiovascular disease (ASCVD), indicators of high ASCVD risk, established kidney disease, or heart failure.

VITAMIN D3:

This section focuses on seven diseases, conditions, and interventions in which vitamin D might be involved: bone health and osteoporosis, cancer, cardiovascular disease (CVD), depression, multiple sclerosis (MS), type 2 diabetes, and weight loss.

Among postmenopausal women and older men, many clinical trials have shown that supplements of both vitamin D and calcium result in small increases in bone mineral density throughout the skeleton. They also help reduce fracture rates in institutionalized older people.

Laboratory and animal studies suggest that vitamin D might inhibit carcinogenesis and slow tumor progression by, for example, promoting cell differentiation and inhibiting metastasis. Vitamin D might also have anti-inflammatory, immunomodulatory, proapoptotic, and antiangiogenic effects. Observational studies and clinical trials provide mixed evidence on whether vitamin D intakes or serum levels affect cancer incidence, progression, or mortality risk.

Vitamin D helps regulate the renin-angiotensin-aldosterone system (and thereby blood pressure), vascular cell growth, and inflammatory and fibrotic pathways. Vitamin D deficiency is associated with vascular dysfunction, arterial stiffening, left ventricular hypertrophy, and hyperlipidemia. For these reasons, vitamin D has been linked to heart health and risk of CVD.

Vitamin D is involved in various brain processes, and vitamin D receptors are present on neurons and glia in areas of the brain thought to be involved in the pathophysiology of depression.

Many epidemiological and genetic studies have shown an association between Multiple Sclerosis (MS) and low 25(OH)D levels before and after the disease begins. Observational studies suggest that adequate vitamin D levels might reduce the risk of contracting MS and, once MS is present, decrease the risk of relapse and slow the disease's progression.

Vitamin D plays a role in glucose metabolism. It stimulates insulin secretion via the vitamin D receptor on pancreatic beta cells and reduces peripheral insulin resistance through vitamin D receptors in the muscles and liver. Vitamin D might be involved in the pathophysiology of type 2 diabetes through its effects on glucose metabolism and insulin signaling as well as its ability to reduce inflammation and improve pancreatic beta-cell function.

Low vitamin D status appears to be associated with type 2 diabetes and most other insulin resistance disorders reported to date.In persons with prediabetes, vitamin D supplementation reduces the risk of T2DM and increases the reversion rate of prediabetes to normoglycemia. The benefit of the prevention of T2DM could be limited to nonobese subjects.

Moreover, Vitamin D, among many benefits, has positive outcomes on hemoglobin A1c (HbA1c) control. It aids in insulin secretion and sensitivity. The clinical significance of Vitamin D administration in DM II from a glucose homeostasis perspective, and complications such as nephropathy, neuropathy, and retinopathy. Vitamin D had a clinical positive impact on glucose level, particularly on hemoglobin A1c (HbA1c) reduction, alleviation of diabetic neuropathy and nephropathy symptoms, and hyperglycemia induced oxidative stress on the retinal cells.

Observational studies indicate that greater body weights are associated with lower vitamin D status, and obese individuals frequently have marginal or deficient circulating 25(OH)D levels.

VITAMIN K2:

Type 2 diabetic patients are at high risk of bone fractures even if their bone mineral density is normal or high. This is likely explained by poor bone quality and extraskeletal factors. Vitamin K(2) stimulates γ-carboxylation of osteocalcin and can increase bone formation through steroid and xenobiotic receptors. study showed that vitamin K(2) administration in a type 2 diabetic had the following skeletal benefits: increased serum osteocalcin, improved collagen cross-link profiles, and increased bone strength. These new findings suggesting a possible beneficial effect of vitamin K(2) supplementation on bone quality in type 2 diabetes.

Micronutrients are gaining acceptance as an important nutritional therapy for the prevention and/or management of diabetes and its associated health risks. Although a very small quantity of micronutrients are required for specific functions in our bodies, moderate deficiencies can lead to serious health issues. Impaired insulin sensitivity and glucose intolerance play a major role in the development of diabetic pathophysiology. Vitamin K is well known for its function in blood coagulation. Moreover, several human studies reported the beneficial role of vitamin K supplementation in improving insulin sensitivity and glucose tolerance, preventing insulin resistance, and reducing the risk of type 2 diabetes (T2 D). Both animal and human studies have suggested that vitamin K-dependent protein (osteocalcin [OC]), regulation of adipokine levels, antiinflammatory properties, and lipid-lowering effects may mediate the beneficial function of vitamin K in insulin sensitivity and glucose tolerance.

Studies showed vitamin K2 intake reduced 7% T2DM risk with each 10-μg increment.

* Vitamin K2 has a more significant effect than vitamin K1 on T2DM.
* Vitamin K2 increased insulin sensitivity via osteocalcin metabolism.

  . Vitamin K2 improved IR via anti-inflammatory property and lipid-lowering effects.
* Vitamin K2 suppresses inflammation via inactivating NF-κB signalling pathway.
* Vitamin K2 supplementation decreases fat accumulation and serum triglycerides.

An important strategy for controlling T2DM is the use of vitamin supplements. vitamin K supplementation can effectively improve clinical features of diabetes. Vitamin K has different forms, including vitamin K1 (phylloquinone), vitamin K2 (menaquinone or MK) and vitamin K3 (synthetic form named menadione). Differences in the chemical structure of K1 (phylloquinone) and K2 (menaquinone) have led to differences in their uptake and bioavailability. Adsorption, bioavailability and the half-life of K2 is higher than K1. Another study suggested that vitamin K supplementation in T2DM results in improved glycemic status, including: FBS, HbA1C, FI and HOMA-IR. Vitamin K supplementation may also help with body weight maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40-60 years
* Type 2 DM for at least 10 years
* Currently on at least 1 regular monotherapy of oral Anti-hyperglycemic agents
* Vitamin D levels < 30 mg/mL

Exclusion Criteria:

Other types of Diabetes

• Pregnant or lactating mothers or women of child bearing potential not practicing an acceptable method of birth control

Diabetic ketoacidosis (DKA) and/or recent history of DKA in last 3 months

* Severe renal (CKD Stage 5, ESRD, eGFR < 45 mL/min/1.73 m 2 or dialysis) or hepatic impairment (Liver cirrhosis, hepatitis)
* Presence of any of the following diseases o Hypothyroidism/hyperthyroidism o Blood disorders causing unstable red blood cells or hemolysis, blood dyscrasias o Benign Prostate Hyperplasia o Recent Acute Coronary Syndrome (ACS), stroke or transient Ischemic attack (TIA) in last 3 months.
* Patients taking any of the following medications o Anti-epileptics o Diuretics o Insulin or Insulin Secretagogues o Anti-Obesity or weight loss drugs (eg Orlistat)
* Presence of any granulomatous disease like Tuberculosis or sarcoidosis
* History of allergy or hypersensitivity reaction to Empagliflozin, Cholecalciferol or Menaquinone MK-7
* Risk of hypotension including low systolic Blood pressure
* Patients with recurrent and/or recent (past 3 months) history of Urosepsis, Pyelonephritis, Urinary Tract Infections and genital mycotic infections and/or positive Urine Culture
* High Low Density Lipoprotein (LDL-C) > 160 mg/dL

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 340 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 3 months
  Mean change in HbA1c levels in % from baseline to end of study at 3 months
Fasting Blood Sugar (FBS) | 3 months
  Mean change in Fasting blood sugar ( serum levels of Glucose in mg/dL after 6-8 hours of fasting) from baseline to end of study at 3 months
Random Blood Sugar (RBS) | 3 months
  Mean change in Random blood sugar from baseline to end of study at 3 months. ( A random glucose test is one method for measuring the amount of glucose or sugar circulating in a person's blood. Doctors perform this test and use the result to determine whether a person is likely to have diabetes)
Hypotension | 3 months
  Number of times ( frequency) the patient experienced low blood pressure during the defined study time frame
Dehydration | 3 months
  Number of times (frequency) the patient felt dehydrated during the defined time frame
Urinary Tract Infection | 3 months
  Incidence of clinically diagnosed or patient's self-reported Urinary Tract Infections
Diabetic Ketoacidosis | 3 months
  Incidence of clinically diagnosed Diabetic Ketoacidosis during the defined time frame of study
Fungal infections | 3 months
  Incidence of clinically diagnosed or patient's self-reported Fungal Infections during the time frame of study
Mean change on body weight in kilogram (kg) | 3 months
  Mean change in body weight in kilograms during the defined study time frame of 3 months from baseline
Blood Pressure change | 3 months
  Mean Change in Systolic and Diastolic blood pressures at baseline and at the end of the study
Total Cholesterol | 3 months
  Mean Change in Total Cholesterol at baseline and at the end of the study
High Density Lipoprotein (HDL) | 3 months
  Mean Change in High Density Lipoprotein (HDL) at baseline and at the end of the study
Low Density Lipoprotein (LDL-C) | 3 months
  Mean Change in Low Density Lipoprotein (LDL) at baseline and at the end of the study
Triglycerides | 3 months
  Mean Change in Triglycerides at baseline and at the end of the study

SECONDARY OUTCOMES:
Pain Visual Analogue Scale (VAS) | 3 months
  Mean Change in Pain Visual Analogue Scale (VAS) at baseline and at the end of the study. The visual analog scale (VAS) is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 100 mm horizontal line, and this rating is then measured from the left edge (=VAS score). Higher the score, more the pain.
Weakness/fatigue | 3 months
  Patient's reported weakness, fatigue, tiredness or any subjective improvement
Muscular aches and pain | 3 months
  Presence/absence of muscular aches and pain
Backache | 3 months
  Presence/absence of backache and its severity and frequency
Quality of sleep | 3 months
  Patient-reported quality of sleep during the study period
Mood swings | 3 months
  Patient-reported incidence/frequency of mood swings including episodes of depression and anxiety
Satisfaction with treatment and life | 3 months
  Patient-reported overall satisfaction with treatment and life

CONTACTS AND LOCATIONS:
Overall Officials: Javed Akram, MRCP,FRCP, Study Chair — University of Health Sciences Lahore; Zaman Shaikh, MRCP,MSc, Principal Investigator — Sir Syed Medical hospital, Khi College of Sciences & Qayyumabad,Khi
Locations (1):
- University of Health Sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wanner C, Inzucchi SE, Lachin JM, Fitchett D, von Eynatten M, Mattheus M, Johansen OE, Woerle HJ, Broedl UC, Zinman B; EMPA-REG OUTCOME Investigators. Empagliflozin and Progression of Kidney Disease in Type 2 Diabetes. N Engl J Med. 2016 Jul 28;375(4):323-34. doi: 10.1056/NEJMoa1515920. Epub 2016 Jun 14. PMID 27299675